CLINICAL TRIAL: NCT04090385
Title: Multifocal Neuromodulation in Motor and Cognitive Function of People With Parkinson's Disease: Randomized Controlled Trial
Brief Title: Multifocal Neuromodulation in Motor and Cognitive Function of People With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Principal Investigator and Professor, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NeuroPark
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS over M1 and DLPFC (Experimental): Anodic transcranial direct current stimulation (tDCS) over left primary motor cortex (M1) and left dorsolateral prefrontal cortex (DLPFC). Duration: 20 minutes; Intensity: 2mA.
  Interventions: Device: Transcranial Direct Current Stimulation
- tDCS over M1 and FPA (Experimental): Anodic transcranial direct current stimulation (tDCS) over left primary motor cortex (M1) and left frontal polar area (FPA). Duration: 20 minutes; Intensity: 2mA.
  Interventions: Device: Transcranial Direct Current Stimulation
- tDCS over M1 (Active Comparator): Anodic transcranial direct current stimulation (tDCS) over left primary motor cortex (M1). Duration: 20 minutes; Intensity: 2mA.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Participants will receive 15 sessions of Transcranial Direct Current Stimulation (tDCS) for 20 minutes each at 2 mA intensity, 5 times a week. The current will be delivered via saline-embedded sponge surface electrodes using a battery-powered neurostimulator (TCT-Research, Trans Cranial Technologies, Hong Kong). A small active specific electrode (5x5 cm) will be used to prevent coverage of adjacent areas, resulting in a current density of 0.08 mA / cm². These parameters are within the safe limits established in previous human studies.
  Other Names: tDCS

SUMMARY:
People with Parkinson's disease (PD) experience various motor and nonmotor symptoms throughout its evolution. It is characterized mainly by the presence of tremor, stiffness, bradykinesia and postural instability, leading to progressive functional limitation and impairment in the performance of usual activities of daily living. In addition, patients may have cognitive disorders, memory deficits, problems related to visuospatial dysfunction, difficulties in performing sequential or repetitive movements, freezing, and slow psychological responses. Previous studies analyzed by systematic reviews suggest the efficacy of Transcranial Direct Current Stimulation (tDCS) to improve the motor and non-motor symptoms of PD, depending on the area of stimulation. However, most of these focus only on one specific area. Therefore, the overall objective of this study is to investigate the effects of multifocal neuromodulation on the motor and cognitive function of people with Parkinson's disease.

DETAILED DESCRIPTION:
For this, a randomized, triple-blind clinical trial will be conducted with 60 people with PD, recruited from the reference centers in neurology and physiotherapy in João Pessoa. After recruitment of participants, they will be randomized into three groups: Group 1 - tDCS over Primary motor cortex (M1) + Dorsolateral prefrontal cortex (DLPFC); Group 2 - tDCS over Primary motor cortex + Frontal polar area (FPA); Group 3 - tDCS over Primary motor cortex. In each condition, an initial baseline assessment (T0) will be performed after 15 treatment sessions (T1) and 30 days after the end of the protocol (Follow-up Assessment - T2), during which time participants will not receive any type of treatment. The outcomes evaluated will be: Motor and cognitive function, executive functions, attention and planning, balance, gait speed an quality of life. For all analyzes, the statistical software SPSS (SPSS Inc, Chicago IL, USA) for Windows, version 20.0, will be used and considered significant, an alpha value of 5% (p <0.05 ).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD, issued by a neurologist specializing in movement disorders;
* Disease staging between I and III, according to the modified Hoehn and Yahr scale;
* Be using antiparkinsonian medication regularly;
* Score higher than 24 or 18 (for participants with low education), verified through the Mini Mental State Examination.

Exclusion Criteria:

* Diagnosis of atypical parkinsonism;
* Neurological comorbidities;
* History of epilepsy, neurosurgery (including metal clip implantation) and pacemaker implantation;
* Previous surgical intervention for PD (DBS implantation - deep brain stimulation);
* Presence of severe freezing episodes.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Changes in motor function assessed by the Unified Parkinson's Disease Rating Scale - Part III (UPDRS - III) | Baseline, after 6 weeks, and after 10 weeks (follow-up)
  For this outcome, the Unified Parkinson's Disease Rating Scale - Part III will be used. Section III provides an overall score for movement-related functions and activities (tremor, stiffness, gait, alternating movements, among others). This section is made up of 33 items, which can range from zero (normal) to four (severe), with responses that are linked to commonly accepted clinical terms. The higher the score, the greater the impairment of motor function.
Changes in cognitive function assessed by the Montreal Cognitive Assessment (MoCA) | Baseline, after 6 weeks, and after 10 weeks (follow-up)
  The Montreal Cognitive Assessment (MoCA) is a cognitive screening tool. MoCA is composed of eight cognitive domains, which are scored within a range of 0 to 30 points (higher scores indicate better function): short-term memory; visuospatial skills; executive function; verbal fluency; attention, concentration and working memory; language; sentence repetition; and spatiotemporal orientation.

SECONDARY OUTCOMES:
Changes in attention and mental flexibility assessed by the Trail Making Test - A and B | Baseline, after 6 weeks, and after 10 weeks (follow-up)
  To assess this outcome, the Trail Making Test - Parts A and B will be used. In condition A, the participant must draw lines, without removing the pencil from the paper, to connect numbers in a sequence. In condition B, the participant must draw lines to connect numbers and letters in an alternating numeric and alphabetic sequence. Prior to the execution of the task, a short "training sheet" is presented from both parts, in which the above instructions are given. The final score represents the total time to finish the task execution. When the participant makes a mistake during the test, the examiner should point out the error at the time of the test and ask the examiner to return to the previous circle and continue the test. Thus, errors are not logged, but result in an increase in total time.
Changes in executive functions and planning assessed by the London Tower Task | Baseline, after 6 weeks, and after 10 weeks (follow-up)
  The Tower of London task is very sensitive to evaluate executive dysfunction in PD patients. The Tower of London is made up of three vertical pins of different heights and three colored spheres, with a hole in the center for the pins to fit. The goal is to move them to reproduce, in a given number of moves, the position of a presented target figure. There are 15 problems with increasing difficulty and reduced possibilities for moving parts. Three attempts to resolve the issue are allowed. Will be evaluated: total and average execution time, and total score, obtained by the sum of the points of each step, ranging from 0 to 3.
Changes in working memory assessed by the Digit Span Forward and Backward Test | Baseline, after 6 weeks, and after 10 weeks (follow-up)
  The Digit Span Forward (DSF) is related to the efficiency of attention, while the Digit Span Backward (DSB), the performance of working memory. Both tests involve six pairs of random numeric sequences that the examiner reads aloud at the rate of one per second. During the DSF the participant will have to repeat each sequence of numbers exactly as they were given, while in the DSB they have to repeat each sequence of numbers in the reverse order. When a sequence is repeated correctly, the examiner reads the next one continuing until the subject fails in a set of sequences or repeats the highest sequence correctly. For each digit repeated correctly, one point is given.
Changes in balance assessed by the Mini-BESTest | Baseline, after 6 weeks, and after 10 weeks (follow-up)
  The Mini-BESTest test will be used to evaluate static and dynamic balance in 14 activities. These include TUG (Timed Up and Go), Push and Release Test and gait quality while changing speed, handling obstacles and turning on your own body axis. Each of the 14 items is scored from 0 to 2, with 0 indicating the lowest level of functionality.
Changes in gait speed assessed by 10 Meter Walk Test | Baseline, after 6 weeks, and after 10 weeks (follow-up)
  To evaluate gait speed and cadence will be used the 10 Meter Walk Test (10MWT). A distance of 10 meters will be determined, with 2 meters of initial acceleration and 2 meters for deceleration. Participants will have 3 attempts to travel the distance, walking as fast as possible without running. An average of the time spent during the three attempts will be calculated. Finally, the number of steps will be counted by visual observation.
Changes in quality of life for people with Parkinson's disease assessed by the Parkinson's Disease Questionnaire (PDQ-39) | Baseline, after 6 weeks, and after 10 weeks (follow-up)
  PDQ-39 is a specific quality of life assessment scale for Parkinson's disease and comprises 39 items that can be answered with five different response options: "never"; "Sometimes"; "sometimes"; "often"; "Always" or "it's impossible for me". The instrument is divided into eight dimensions: Mobility (10 items), Daily Living Activities (6 items), Emotional Wellbeing (6 items), Stigma (4 items), Social Support (3 items), Cognition (4 items) , Communication (3 items) and Body Discomfort (3 items). The total score for each individual is calculated according to the following formula: 100 x (sum of patient scores on 39 questions / 4 x 39). The score of each dimension is obtained in the same way as the total score. A low score indicates better perception of quality of life by the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, Principal Investigator — Federal University of Paraiba
Locations (1):
- Suellen Marinho Andrade, João Pessoa, Paraíba, Brazil